CLINICAL TRIAL: NCT07383714
Title: Nudging Parental Action With A Randomized Controlled Trial of Text Messaging Intervention for Suicide Prevention
Brief Title: Nudging Parental Actions for Youth Suicide Prevention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The Texas Child Mental Health Care Consortium (TCMHCC) (Unknown)
Responsible Party: Principal Investigator, Rabia Ayvaci, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU20252399; GAA202508-0021 (Other Grant/Funding Number: New and Emerging Children's Mental Health Researchers Initiative)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Suicide; Suicide Attempt
Keywords: suicide; digital health; lethal means restriction
MeSH Terms: conditions — Suicide; Suicide, Attempted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The person analyzing the data will be blinded to group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (No Intervention): Treatment as usual (ED-based lethal means counseling)
- Direct Nudge (Active Comparator): Thrice-weekly direct text messages encouraging Lethal Mean Restriction practices.
  Interventions: Other: Text-messaging for safety reminders
- Risk-Framing Nudge Arm (Experimental): Thrice-weekly direct text messages encouraging Lethal Mean Restriction practices and suicide risk statistics to recalibrate parental risk perception
  Interventions: Other: Text-messaging with safety reminders and risk framing

INTERVENTIONS:
Other: Text-messaging for safety reminders — The intervention consists of thrice-weekly, behaviorally informed text messages delivered to parents over six weeks period.
  Arms: Direct Nudge
Other: Text-messaging with safety reminders and risk framing — Thrice-weekly messages incorporating safety precautions and evidence-based suicide risk statistics to recalibrate parental risk perception.
  Arms: Risk-Framing Nudge Arm

SUMMARY:
The goal of the study is to determine effectiveness of a behaviorally informed text messaging intervention to help parents increase safety practices and reduce their teens' access to lethal means following a suicide-related emergency department visit.

DETAILED DESCRIPTION:
This study tests a text messaging program that helps parents keep their teens safe after a visit to the emergency department for suicidal thoughts or behavior. Adolescents face a higher risk of suicide after leaving the emergency department, and limiting access to lethal means such as firearms, medications, or other dangerous items can help prevent suicide. The investigators invite parents and their teens aged 12 to 17 who visit the emergency department at Children's Medical Center Dallas for suicide-related reasons to join the study. After enrolling, families will be randomly assigned to one of three groups. The first group receives usual care, which includes standard counseling about keeping teens safe in the emergency room and no study text messages. The second group receives direct text messages three times a week with reminders about safety reminders. The third group receives risk-framing text messages three times a week, which include safety reminders and information about suicide risk following an emergency room visit to motivate parents to take action. The study measures whether these text messages help parents follow safety recommendations at home. Parents and teens complete short surveys at the start of the study, six weeks later, and twelve weeks later. The study also tracks whether the teen returns to the emergency department or attempts suicide again. The study aims to determine if text messages can increase parental safety practices, reduce teens' access to lethal means, and prevent future suicide attempts. UT Southwestern Medical Center and Children's Health Dallas conduct the study. Messages are delivered through a secure, HIPAA-compliant virtual platform to ensure privacy.

ELIGIBILITY:
Inclusion Criteria:

* Guardian must be able and willing to provide informed consent, and the participant must be able and willing to provide assent.
* Parent and adolescent willingness and ability to participate in study procedures and complete assessments at baseline, 6 weeks, and 12 weeks.
* Presentation to the ED for a suicide-related emergency, defined as suicidal ideation within the last 2 weeks or a suicide attempt within the past month.
* Adolescents aged 12-17 years during the consent.
* Access to a mobile phone with text messaging capability for the parent/legal guardian.
* Ability to communicate in English.

Exclusion Criteria:

* Absence of a legal guardian capable of providing consent.
* Parents/legal guardians without access to a mobile phone with texting capability.
* Inability to communicate in English.
* Adolescents in state custody or under legal restrictions that prevent study participation.
* Adolescents involved in the justice system in a manner that would interfere with study participation.
* Adolescents with autism spectrum disorder or intellectual development disorder needing substantial or very substantial support

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Parent-reported adherence to lethal means restriction (LMR) | Baseline to 6 weeks
  Change in parental adherence to lethal means restriction practices will be assessed using the Parent Adherence to Lethal Means Restriction (PA-LMR), a structured parent-report survey measuring adherence to multiple lethal means restriction behaviors. Items are rated on a Likert scale, with total scores ranging from 11 to 55; higher scores indicate greater adherence.

SECONDARY OUTCOMES:
Adolescent Perceived Access to Lethal Means | Baseline to 6 weeks
  Perceived Access to Lethal Means is a self-report measure assessing adolescents' perceptions of their access to potentially lethal methods. Items assess the perceived ease of access, with total scores ranging from 5 to 30; higher scores indicate greater perceived access to lethal means.

OTHER OUTCOMES:
Exploratory Outcome | Baseline to 12 weeks
  Number of participants (adolescents) with a suicide-related Emergency Department revisit and/or suicide attempt within 12 weeks post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Emine Rabia Ayvaci, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No
No individual participant data is planned to be shared with other researchers.

REFERENCES:
- [Background] Tversky A, Kahneman D. The framing of decisions and the psychology of choice. Science. 1981 Jan 30;211(4481):453-8. doi: 10.1126/science.7455683.
- [Background] Bauer BW, Capron DW. How Behavioral Economics and Nudges Could Help Diminish Irrationality in Suicide-Related Decisions. Perspect Psychol Sci. 2020 Jan;15(1):44-61. doi: 10.1177/1745691619866463. Epub 2019 Nov 7. PMID 31697611
- [Background] Barber CW, Miller MJ. Reducing a suicidal person's access to lethal means of suicide: a research agenda. Am J Prev Med. 2014 Sep;47(3 Suppl 2):S264-72. doi: 10.1016/j.amepre.2014.05.028. PMID 25145749